CLINICAL TRIAL: NCT07399691
Title: Effect of Adding Dexamethasone to Bupivacaine in Ultrasound-Guided Supraclavicular Brachial Plexus Blocks Versus Bupivacaine Alone for Upper Limb Orthopaedic Surgery
Acronym: SCBPBs
Status: Completed | Type: Observational
Sponsor: Arsi University (Other)
Responsible Party: Principal Investigator, Mohammed Gebi, lecturer at arsi university, Arsi University
Other Study IDs: No-A/CHS/RC/19/2023
Record Dates: First submitted 2026-01-23; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Dexamethasone; Bupivacaine; Upper Limb Surgery
Keywords: dexamethasone,Bupivacaine,Analgesia,supraclavicular block
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group DB: Patients received a supraclavicular brachial plexus block with dexamethasone 2 ml (8 mg) added to 38 ml of 0.25 % bupivacaine.
  Interventions: Drug: Dexamethasone 8 mg
- Group B: Patients received a supraclavicular brachial plexus block with 40 ml of 0.25 % bupivacaine alone.

INTERVENTIONS:
Drug: Dexamethasone 8 mg — Adding 8 mg of dexamethasone to bupivacaine for ultrasound-guided supraclavicular block
  Groups: Group DB

SUMMARY:
* SCBPBs provides optimal conditions for procedures performed below the mid-upper arm (elbow, forearm, wrist, hand) due to its high success rate and ease of access.
* Dexamethasone, when administered perineurally as an adjuvant for a supraclavicular block, demonstrated early onset of sensory and motor block, a prolonged duration of sensory and motor block, and a lower number of rescue analgesics as compared to bupivacaine alone.
* A combination of dexamethasone and bupivacaine is paramount in adult orthopeadic patient to enhance the efficacy of pain management under ultrasound-guided supraclavicular brachial plexus block.

ELIGIBILITY:
Inclusion Criteria:

Aged 18-60 years with ASA I and II who were scheduled for elective elbow, forearm, or hand surgery under ultrasound-guided supraclavicular block.

Exclusion Criteria:

Patients who refused, used local anaesthetics other than bupivacaine, had multiple traumas, addition of another additive, bleeding disorders, patients diagnosed with chronic pain, cancer pain, local infection at the injection site, history of local anaesthetic allergy, patients with anxiety, and inability to comprehend or use the pain rating scale

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study included 54 patients aged 18-60 years with ASA I and II who were scheduled for elective elbow, forearm, or hand surgery under ultrasound-guided supraclavicular bloc
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
The onset of sensory and motor blockade, and the duration of sensory and motor blockade in minutes. | with in the first 24hrs after procedure
  1. The onset of sensory: the period between injecting a study solution and losing sensation to a pinprick at every nerve distribution
  2. The onset of motor block: The duration between the injection of the study solution and paresis in every nerve distribution.
  3. duration of sensory: the period between the onset of a sensory block and the complete restoration of sensation.
  4. Duration of motor block: the period between the onset of a motor block and the complete restoration of motor function.

SECONDARY OUTCOMES:
postoperative pain score by a visual analogue scale | with in the first 24 hrs after procedure
  This assesses behavioural or subjective phenomena by having the participant choose an alternative from a gradient ranging from 0 = (no pain) to 100 = worst possible pain. Based on the VAS score, 0-20 mm = no pain; 21-40 mm = mild pain; 41-60 mm = moderate pain; 61-80 mm = severe pain; and 81-100 mm = the worst pain imaginable
First analgesic request time | With in the first 24 hrs after surgery
  The first postoperative period, when patients require pain treatment if the visual analogue score is>4

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammed Gebi, Āsela, Ethiopia

IPD SHARING:
Plan to Share IPD: No